CLINICAL TRIAL: NCT07122297
Title: Clinical Evaluation of Different Gingival Displacement Methods
Brief Title: Evaluation of Gingival Displacement Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, GAYE SAĞLAM, Associate Professor, Zonguldak Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015/121
Record Dates: First submitted 2025-07-24; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Gingival Displacement
Keywords: Cord, Diode laser, Paste, Retraction
MeSH Terms: conditions — Cone-Rod Dystrophies | interventions — Lasers, Semiconductor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group K (Experimental): Retraction cord impregnated with 15% ferric sulfate is used for gingival displacement
  Interventions: Procedure: Retraction cord
- Group P1 (Experimental): A retraction paste in capsule form, containing 15% aluminum chloride is used for gingival displacement.
  Interventions: Procedure: Retraction paste in capsule form
- Group P2 (Experimental): A retraction paste in injector form is used for gingival displacement.
  Interventions: Procedure: Retraction paste in injector form
- Group L (Experimental): A diode laser is used for gingival displacement.
  Interventions: Procedure: Diode Laser

INTERVENTIONS:
Procedure: Retraction cord — A thin cord (type "00") was soaked in 15% ferric sulfate ferric sulfate hemostatic solution and carefully packed into the gingival sulcus. After 3 minutes, the cord was removed and the sulcus was rinsed. This is a traditional mechanical gingival displacement method.
  Arms: Group K
Procedure: Retraction paste in capsule form — A retraction paste was applied using a capsule tip placed around the gingival margin. The paste remained in place for 3 minutes and was then rinsed off with air-water spray. This is a non-traumatic chemical displacement technique.
  Arms: Group P1
Procedure: Retraction paste in injector form — Retractrion paste in injector form with compression cap (15% aluminum chloride) was injected into the sulcus, and a cotton compression cap was placed over the tooth. Patients gently bit on the cap for 3 minutes to apply pressure. Afterward, the paste and cap were removed and the area was rinsed. This method combines chemical and slight mechanical displacement.
  Arms: Group P2
Procedure: Diode Laser — A 810-nm diode laser with a 400-micron fiber optic tip was used in contact mode to ablate the sulcular epithelium. The laser was operated at 1.0 W with pulsed settings. The procedure was completed by wiping the area with saline to remove residues. This technique enables precise, bloodless gingival retraction with minimal trauma.
  Arms: Group L

SUMMARY:
This clinical study is being conducted to compare four different methods used to temporarily push the gums away from the teeth during dental procedures. This process, called gingival displacement, is important for dentists to clearly see and work around the tooth when placing crowns or taking impressions. The four methods being studied include: A retraction cord soaked in a special solution, A retraction paste in a capsule, A retraction paste applied with a cap, A soft tissue laser (called a diode laser). Each method is applied to teeth that need crown treatment. The goal is to find out which method moves the gum tissue the most effectively, and which one causes the least bleeding. Fifty-two teeth in total were treated using one of these four methods. Before and after treatment, gum measurements were taken to evaluate how much the gums moved and how much bleeding occurred. By studying these methods, the researchers hope to help dentists choose the most effective and least invasive technique for each patient's needs.

DETAILED DESCRIPTION:
This study was designed to compare four different gingival displacement techniques in terms of their effectiveness in achieving both vertical and horizontal gingival retraction. The aim was to evaluate the extent of gingival tissue displacement and the associated clinical outcomes, such as bleeding, for each intervention, thereby helping clinicians select the most appropriate method in various clinical scenarios.

Systemically healthy individuals over 18 years of age requiring fixed prosthodontic treatment with abutment teeth in the canine, premolar, or molar regions were included in this study. Fifty-two teeth were randomly assigned to four groups (n=13) and prepared with an epigingival margin and chamfer finish line.

Group K: 15% ferric sulfate-impregnated retraction cord Group P1: Retraction paste in capsule form containing 15% aluminum chloride Group P2: Retraction paste in injector form containing 15% aluminum chloride with a compression cap Group L: 810-nm diode laser All teeth were prepared with an epigingival margin and chamfer finish line to standardize clinical conditions. Gingival displacement was evaluated in two dimensions: Vertical displacement was measured using a periodontal probe before and one week after gingival displacement. Horizontal displacement was assessed by taking polyvinyl siloxane impressions at the same time points. These impressions were analyzed under a stereomicroscope, and displacement was quantified using calibrated image analysis software.

Each intervention was applied following standardized protocols: In Groups K, P1, and P2, materials were applied for 3 minutes. In Group L, the diode laser was used in contact mode to ablate the sulcular epithelium using specific pulse and power settings (1.0 W, 1 ms pulse length). In addition to displacement measurements, post-displacement hemorrhage was clinically evaluated as a secondary outcome to assess tissue trauma and hemostatic effectiveness. All clinical procedures and measurements were performed by the same calibrated operator to ensure consistency.

Statistical analysis was conducted using SPSS software. The distribution of data was tested with the Shapiro-Wilk test. Inter-group comparisons were analyzed with the Kruskal-Wallis and Dunn's post hoc tests; intra-group comparisons used paired t-tests or Wilcoxon Signed Rank tests, depending on data distribution. A p-value < 0.05 was considered statistically significant.

The results are intended to guide clinicians in selecting gingival displacement techniques based on quantitative performance and clinical behavior under standardized conditions.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age
* Having clinically and radiographically healthy periodontal tissues (probing depth not exceeding 3 mm, no bleeding on probing, no gingival recession, no bone loss)
* Having completed Phase I periodontal therapy
* Having no systemic disease that could affect periodontal health
* Having abutment teeth located in the canine, premolar, or molar regions
* Absence of any developmental anomalies in the abutment teeth
* Absence of age-related degenerative changes in the abutment teeth

Exclusion Criteria:

* Being under 18 years of age
* Having an uncontrolled or periodontal-health-affecting systemic disease
* Not having periodontally healthy tissues
* Having adjacent abutment teeth
* Having previously prepared abutment teeth
* Presence of any developmental anomaly in the abutment teeth
* Presence of age-related degenerative changes in the abutment teeth

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Horizontal Gingival Displacement | Baseline and 1 week post-displacement
  The amount of tissue movement away from the tooth surface (laterally). Measured by comparing stereomicroscopic images of polyvinyl siloxane (PVS) impressions taken before and after displacement. The horizontal gap is measured in millimeters.
Vertical Gingival Displacement | Baseline and 1 week post-displacement
  The amount of tissue movement in the vertical direction (apically) after using each gingival displacement method.

SECONDARY OUTCOMES:
Gingival Hemorrhage | Immediately post-displacement
  The amount of bleeding observed after application of the gingival displacement method.
  Gingival hemorrhage was assessed immediately after gingival displacement and removal of the applied materials from the tooth and gingiva. Bleeding was recorded using a score system:
  0 - No bleeding observed
  1. - Bleeding that could be controlled within 1 minute
  2. - Bleeding that could not be controlled within 1 minute

CONTACTS AND LOCATIONS:
Overall Officials: Seda CENGİZ, DDS, Phd, Study Director — Professor, Counsellor for Education of Turkish Embassy in Vienna, Prinz-Eugen, Vienna, Austria.

IPD SHARING:
Plan to Share IPD: No